CLINICAL TRIAL: NCT02682654
Title: A Multi-Site Evaluation of the Pain Relief, Support, Fit and Comfort From Use of a Custom Knee or Ankle Brace in Persons Suffering From Chronic Ankle or Knee Pain and Instability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: 18325
Record Dates: First submitted 2016-02-11; First posted 2016-02-15 (Estimated); Last update posted 2018-12-12 (Actual); Status verified 2018-12

CONDITIONS: Joint Instability
Keywords: Pain; Ankle; Knee; Brace
MeSH Terms: conditions — Joint Instability; Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ankle/Knee brace (Experimental): Dr. Scholl's Prototype Ankle or Knee Brace
  Interventions: Device: Dr. Scholl's Prototype Ankle Brace; Device: Dr. Scholl's Prototype Knee Brace

INTERVENTIONS:
Device: Dr. Scholl's Prototype Ankle Brace — Subjects will be instructed to wear the assigned Ankle/Knee brace for 8 ± 2 hours per day, for a minimun of 5 days out of a 7-day/1 week wear period.
Device: Dr. Scholl's Prototype Knee Brace — Subjects will be instructed to wear the assigned Ankle/Knee brace for 8 ± 2 hours per day, for a minimun of 5 days out of a 7-day/1 week wear period.

SUMMARY:
This study will look to examine the overall performance of a custom fit knee or ankle brace as a means of providing ankle or knee joint support in subjects that have determined the need for bracing based upon chronic joint instability and/or joint swelling and pain following daily activity.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must indicate that they currently have weakened ankles or knees and that they experience chronic discomfort after performing daily activities.
* Subjects must suffer from pain assessed on a 100 mm (10 cm) Visual Analog Scale (VAS) of ≥20 mm to ≤ 90 mm for subjects with either unstable ankle or unstable knee, at Visit 1 and 2.
* Subjects must be able to walk unaided by cane or walker.
* Subjects must not have a noticeable limp or other permanent ailment that interferes with normal gait.
* Subjects free of other types of health problems that, in the opinion of the Investigator, could influence their ability to participate.
* If subjects are taking pain medication (prescription or Over-the-counter (OTC)) for a chronic condition, they may continue that medication as long as they have been on a stable dose for at least 2 months, and agree to continue their regular dose and regimen for the duration of the study.
* Subjects must be willing to undergo a 1-week period without a brace and then willing to wear a brace for a 1-week period, that is: 8 ±2 hours a day for a minimum of 5 out of 7 days.

Exclusion Criteria:

* Subjects with an ankle or knee pain and instability which is due to a recent sprains, strains, or other non-reversible injury to the knee or ankle.
* Subjects who have diabetes, circulatory problems, open wounds, and lack of sensation in the ankles, knees, or feet or any problems that would make brace wear uncomfortable or inappropriate.
* Subjects who wear a physician-prescribed orthotic device, prescription shoes or back braces.
* Subjects who are undergoing traction or manipulative back adjustments or have had a traumatic injury to the lower extremity (deemed of non-overuse nature), which in the opinion of the examining Investigator would interfere with the study evaluations.
* Subjects whose condition requires surgery or other medical intervention or who have undergone foot back or knee surgery within the past 3 months or with any planned surgeries and/or invasive medical procedures during the course of the study.
* Subjects who are currently taking an opioid based pain medication or have taken such medication within 2 months prior to Visit 1.
* Subjects who are taking any chronic pain medication (prescription or OTC) for at least 2 months, who do not agree to continue taking it at the same dose and regimen throughout the study.
* Subjects who have severely painful bunions, warts, corns and/or calluses, severely overlapping toes or lesions on the bottom of their foot.
* Subjects who have sensitivities or allergies to plastics or adhesives.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 183 (Actual)
Dates: Start 2016-02-05 (Actual); Primary Completion 2016-04-26 (Actual); Study Completion 2016-04-26 (Actual)

PRIMARY OUTCOMES:
Comfort | Up to 15 days
  Comfort is assessed utilizing a 7-point Comfort/Discomfort Likert scale.
Pain Relief of Knee or Ankle joint | Up to 15 days
  Evaluation of Knee or Ankle joint pain will be performed using the Visual Analog Scale utilizing a 100 mm line defined at each end of the line by 0 = no pain and 100 = Worst pain possible.

SECONDARY OUTCOMES:
Product Fit | Up to 15 days
  Product Fit is assessed utilizing a 7-point scale.
Product Support | Up to 15 days
  Support is assessed utilizing a 5-point scale.
Freedom of Movement | Up to 15 days
  Freedom of Movement is assessed utilizing a 6-point scale.
Subjective Questions | Up to 15 days
  Applicable subjective questions will be assessed utilizing the subjective questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (2):
- United States (2):
  - Colorado Springs, Colorado
  - Richardson, Texas